CLINICAL TRIAL: NCT04533113
Title: Carious Tissue Selective Removal on Permanent Posterior Teeth. A Randomized Controlled Clinical Study.
Brief Title: Carious Tissue Selective Removal on Permanent Posterior Teeth.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Juan Gonzalo Olivieri (Other)
Responsible Party: Sponsor-Investigator, Juan Gonzalo Olivieri, Principal investigator, Universitat Internacional de Catalunya
Organization: Universitat Internacional de Catalunya (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDECL201804
Record Dates: First submitted 2020-08-27; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Dental Caries; Dental Materials
Keywords: Dental caries; Dental materials; Outcome; Postoperative Pain
MeSH Terms: conditions — Dental Caries; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VitreBond LC (Experimental): VitreBond LC used as a liner after selective carious tissue removal.
  Interventions: Procedure: Carious tissue selective removal
- Biodentine (Experimental): Biodentine used as a liner after selective carious tissue removal.
  Interventions: Procedure: Carious tissue selective removal
- Theracal (Experimental): Theracal used as a liner after selective carious tissue removal.
  Interventions: Procedure: Carious tissue selective removal

INTERVENTIONS:
Procedure: Carious tissue selective removal — Carious tissue selective removal in deep carious lesions in posterior teeth, using one of three materials as a liner under the final composite restoration

SUMMARY:
This study is a prospective randomized controlled study of patients who come to the University. The aim is to evaluate the success rate of selective removal of carious tissue in deep lesions of posterior teeth. Three different materials will be used as liners (VitreBond ™Plus, BioDentine™, and Theracal™ LC). Post-operative pain, clinical, and radiographic success will be evaluated at one, two, and five-year follow-up. The null hypothesis is that there will be no statistically significant differences in rates of successful treatment with the three materials used.

ELIGIBILITY:
Inclusion Criteria:

* Patients that demonstrate understanding of the study and willingness to participate as evidenced by signing the voluntary informed consent and received a signed and dated copy of the informed consent form.
* Understands and is willing to comply with all study procedures and restrictions.
* Not presence of clinically significant and relevant abnormalities of clinical history or oral examination.
* Diagnosis of normal pulp or reversible pulpitis.
* No presence of periapical periodontitis
* Posterior teeth

Exclusion Criteria:

General: Patients with systemic diseases, diabetes, immunocompromised and pregnant women, or any clinically significant or relevant oral abnormalities.

Specific: Impossibility of restoration, diagnosis of irreversible pulpitis or necrosis, preoperative pain

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Clinical post-operative pain | Immediately post-treatment
  VAS score of patient' level of pain, from no pain to extreme pain
Clinical post-operative pain | 8 hours post-treatment
  VAS score of patient' level of pain, from no pain to extreme pain
Clinical post-operative pain | 24 hours post-treatment
  VAS score of patient' level of pain, from no pain to extreme pain
Clinical post-operative pain | 48 hours post-treatment
  VAS score of patient' level of pain, from no pain to extreme pain
Clinical signs or symptoms of pulp or periapical disease | 1 year
  Absence/presence of clinical signs or symptoms of pulp or periapical disease
Clinical signs or symptoms of pulp or periapical disease | 2 years
  Absence/presence of clinical signs or symptoms of pulp or periapical disease
Clinical signs or symptoms of pulp or periapical disease | 5 years
  Absence/presence of clinical signs or symptoms of pulp or periapical disease
Radiographic signs of periapical disease | 1 year
  Absence/presence of radiographic apical periodontitis
Radiographic signs of periapical disease | 2 years
  Absence/presence of radiographic apical periodontitis
Radiographic signs of periapical disease | 4 years
  Absence/presence of radiographic apical periodontitis

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No